CLINICAL TRIAL: NCT02271451
Title: Q-collar and Brain Injury Biomarkers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2014-5009
Record Dates: First submitted 2014-10-07; First posted 2014-10-22 (Estimated); Results first posted 2019-09-10 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-08

CONDITIONS: Concussion
Keywords: concussion
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Q collar (Experimental): subjects wearing the q collar
  Interventions: Device: Q collar
- Control (No Intervention): subjects not wearing the Q collar

INTERVENTIONS:
Device: Q collar — collar worn around neck
  Arms: Q collar

SUMMARY:
Significant morbidity, mortality, and related costs are caused by traumatic brain injury (TBI). A simple, effective, and lightweight device worn by athletes or war fighters in the field, designed to mitigate TBI resulting from blast trauma or concussive events, would save lives, and the huge costs currently being experienced for life-treatment of surviving victims. An externally-worn medical device that applies mild jugular compression according to the principle of the Queckenstedt Maneuver (the Device) is being developed by Q30 Labs, LLC (Q30). Initial research suggests that the Device has the potential to reduce the likelihood of TBI. The currently developed collar (Smith 2009; Smith 2011; Smith 2011; Smith 2012) has been approved for studies in humans and the results indicate safety for use during high demand and maximal exertion activities, Study ID: 2013-2240, Institutional Review Board - Federalwide Assurance #00002988). Regarding safety, the externally worn collar is meticulously designed to mimic the body's own omohyoid muscle actions upon the jugular veins that will provide similar pressure and volume increases not to surpass that of a yawn or the mere act of just lying down.

This study will investigate the effectiveness of this device in high school athletes playing a collision or contact sport such as football, hockey, or lacrosse. The high risk sports which utilize helmets during competition will allow for measurements systems to be embedded in the headgear and will not affect play or fit of equipment. Athletes participating in this study will be enrolled into one of two groups 1) device wearing or 2) non-device wearing. By the nature of the sports selected, it is likely this pilot study will primarily include males, however if any female meets inclusion criteria on the team selected they will be included in this pilot investigation. The helmets of all participants will be outfitted with an accelerometer which will measure the magnitude of every impact to the head sustained by the athlete. Effectiveness of the device will be determined by brain imaging during the pre-season, midseason, and end of season time points. A subset of athletes who report a diagnosed concussion will also receive additional brain imaging within the week following the diagnosed concussive event.

DETAILED DESCRIPTION:
The Device has the promise of providing a novel mechanism for reducing or preventing the likelihood of TBI, and may be used in conjunction with other protective equipment. TBI is the leading cause of death in individuals under age 45. The cost of TBI in the U.S. is estimated at anywhere from $50 to $150 billion, annually. The January, 2008 New England Journal of Medicine reports, "Head and neck injuries, including severe brain trauma, have been reported in one quarter of service members who have been evacuated from Iraq and Afghanistan"(Okie 2005; Xydakis 2005; Hoge 2008). The vast majority of these injuries have resulted from exposure to improvised explosive device (IED) blast waves. Head injuries, concussions and the resulting trauma have been in public discussion recently as the National Football League (NFL) deals with a lawsuit regarding head injuries by about one-third of living former NFL players and are also a concern for athletes who participate in a wide range of sports, including hockey, rugby and soccer.

According to NASA, "The oscillation of a fluid caused by an external force, called sloshing, occurs in moving vehicles containing liquid masses, such as trucks, etc." This oscillation occurs when a vessel is only partially filled. Similarly, the brain faces slosh peril during external force impartation. Slosh permits external energies to be absorbed by the contents of a partially filled vessel or container by means of inelastic collisions. Tissues of differing densities can decelerate at different rates creating shear and cavitation. If the collisions between objects or molecules are elastic, the transfer of energies to those objects diminishes, minimizing the energies imparted by slosh.

Woodpeckers, head ramming sheep and all mammals (including mankind) have small, little known and misunderstood muscles in their necks called the omohyoid muscles. Highly G-tolerant creatures of the forest have utilized these muscles to gently restrict outflow of the internal jugular veins thereby "taking up" the excess compliance of the cranial space and ultimately protecting themselves from TBI like tiny "airbags" in a motor vehicle. Rat studies by Smith et al. have demonstrated that the investigators can easily and safely facilitate this muscle's actions by a well-engineered gentle compression over those muscles.

The medical Queckenstedt Maneuver devised to detect spinal cord compression, gently places pressure over the external jugular veins to increase cerebral spinal volume and pressure. In this maneuver, the veins are compressed while a lumber puncture monitors the intracranial pressure. "Normally, the pressure rise to the higher 'plateau' level occurs instantly upon jugular compression to fall again equally fast upon release of the compression"(Gilland 1969). This incredibly simple principle can be employed to protect soldiers and athletes from TBI by safely, and reversibly, increasing intracranial volume and pressure. The neck collar device is made of hytrel (plastic), silicone, metal and fabric that is fitted to the neck providing comfortable and precise jugular compression that potentially mitigates cerebral slosh (Figure 1).

Although the skull, blood, and brain are "almost incompressible," the vasculature tree of the cerebrum is quite reactive and compressible. As volume is added to the cranium, eventually the compensatory reserve volume is surpassed and the intracranial pressure increases slightly. Increasing cerebral blood volume by just 1-3% safely and reversibly reduces compliance of the cerebral vascular tree and diminishes absorption of slosh energies. Jugular compression increases cerebral blood volume almost instantaneously. As mentioned, this degree of increase has significantly mitigated slosh and TBI in laboratory animals and mimics the highly concussion resistant wild animals that are able to reflexively increase cerebral blood volume through jugular compression.

A landmark article, published in the Journal of Neurosurgery, used a standard acceleration-deceleration impact laboratory model of mild TBI. The study showed a successful and marked reduction of axonal injury following Internal Jugular Vein (IJV) compression as indicated by immunohistochemical staining of Amyloid Precursor Proteins (APP) (Smith 2012; Turner 2012). It is argued that IJV compression reduces slosh-mediated brain injury by increasing intracranial blood volume and reducing the compliance and potential for brain movement within the confines of the skull. The potential for such technique to mitigate both linear and rotational brain injury in humans by "internal protection" represents the most novel approach to mitigating TBI.

Summary of Prior Work A. Safety testing in athletes has been approved by the local IRB and was completed in the Cincinnati Children's Hospital Human Performance Laboratory (Study ID: 2013-2240; PI: Gregory Myer). Evaluation of monitored vital signs, biomechanics, cardiorespiratory capacity, postural control, dynamic stabilization, reactive index, concentration and cognition, memory, strength and power in a population of athletes showed no statistically significant adverse effect of wearing a mild jugular vein compressive neck collar compared to a sham arm band.(Myer 2013) Cumulatively, the pre and post safety measures indicate that neurologic parameters of executive function, eye hand coordination, balance, memory and reaction times were unchanged following two hours of physical testing wearing the collar prototype. Acceptance of the compression collar was not different in physiological biomarker response to non-collared condition during maximal oxygen uptake and maximum effort power testing.(Myer 2013) B. Magnetic Resonance Elastography was established at CCHMC in collaboration with The Mayo Clinic to support studies. Under jugular vein compression with the collar, all subjects tolerated the procedure without any untoward effects. The preliminary studies of dynamic shear strain showed no consistent pattern of wave propagation and elasticity, placed upon the vascular and cranial tissues. Analysis of these data continues.

C. Four hundred and ten (410) subjects (ages 12 to 68 years of age) were studied with MEPA (middle ear power analysis) with and without the compression collar and no complaints or untoward effects were noted and no decline in the auditory perception was recorded. The expected changes of reduced Acoustic Reflectance of the inner ear and middle ear (indicative of reduced compliance) were noted only in subgroup analysis of those with jugular vein compression. The results of this study indicate that the neck compression collar prototype may have the potential to safely reduce energy impartation into cranial structures (i.e. the inner ear), however further work is needed with advanced collar designs to establish this effect.

D. fMRI and CO2 reactivity was performed on twelve adults before and after application of jugular vein compression. Results comparing before and after jugular vein compressions (with the collar) yielded no alterations in O2 uptake or glucose metabolism to any portion of the brain.(Fisher 2013)

ELIGIBILITY:
Inclusion Criteria:

* • Normal healthy volunteer

  * Able to provide written consent
  * Must be 14 years or older and a participant on a competitive and organized sports program
  * Neck circumference of 15 ½ - 16 ½ inches

Exclusion Criteria:

* • Unable to provide written consent

  * History of neurological deficits, previous cerebral infarction, or severe head trauma
  * Medical contraindications to restriction of venous outflow via the internal jugular veins (known increased intracerebral pressure, metabolic acidosis or alkalosis)
  * Glaucoma (Narrow Angle or Normal Tension)
  * Hydrocephalus
  * Recent penetrating brain trauma (within 6 months)
  * Known carotid hypersensitivity
  * Known increased intracranial pressure
  * Central vein thrombosis
  * Any known airway obstruction
  * Any known seizure disorder

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2014-10; Primary Completion 2015-05 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory D Myer, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
Overall study results will be presented but individual data will remain de-identified.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Q Collar | Control
Started | 7 | 8
Completed | 7 | 7 (one subject does not have MRI data due to braces)
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Population: One control subject only has EEG data as he has braces and could not do the brain MRI
Groups:
- Total: Total of all reporting groups
Arm/Group | Q Collar | Control | Total
Number analyzed (Participants) | 7 | 8 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7 | 8 | 15
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 7 | 8 | 15
Region of Enrollment [Number; unit: participants]
  United States | 7 | 8 | 15

OUTCOME MEASURES:

1. Primary Outcome: Longitudinal DTI Changes
Description: measured white matter changes, mean diffusivity (MD), and radial diffusivity (RD)
Time Frame: 2 years
Population: Changes seen on DTI imaging
Measure: Mean (Standard Deviation); unit: voxels
Arm/Group | Q Collar | Control
Number analyzed (Participants) | 7 | 7
voxels
  Baseline MD | 0.000809 (0.000056) | 0.000760 (0.000089)
  Mid-Season MD | 0.000763 (0.000072) | 0.000843 (0.000062)
  Baseline RD | 0.000525 (0.000044) | 0.000426 (0.000062)
  Mid-Season RD | 0.000447 (0.000062) | 0.000511 (0.000037)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Q Collar | Control
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/8
Other Adverse Events (participants affected / at risk) | 0/7 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No